CLINICAL TRIAL: NCT05790122
Title: Safety and Efficacy of Sutureless Zero Ischemia Laparoscopic Tumor Enucleation for T1 Stage Renal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: K2023003
Record Dates: First submitted 2023-02-28; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Carcinoma, Renal Cell; Kidney Neoplasms
Keywords: Renal cell carcinoma; Zero ischemia; Unclamped tumor enucleation; Small renal mass; Sutureless
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group PN: The patients undergoing partial nephrectomy.
- Group TE: The patients undergoing renal tumor enucleation.

SUMMARY:
Partial nephrectomy(PN) and tumor enucleation(TE) are the two main methods of Nephron-sparing surgery for early renal cell carcinoma. Because of its blunt separation, TE is often considered to be difficult to completely remove tumor tissue. In addition, compared with PN, TE is more difficult and has higher professional requirements for surgeons. Therefore most surgeons use PN. But Many studies have shown that TE has advantages over PN such as less trauma, faster recovery, and better protection of renal function without increasing the risk of tumor recurrence.

The main renal artery should be clamped during PN to achieve a relatively bloodless operation environment to ensure the safety of tumor resection. However, too long warm ischemia time will inevitably affect the function of normal renal tissue. Studies have shown that shortening the time of renal ischemia is closely related to the recovery of renal function after the operation. So reducing the time of warm ischemia until zero ischemia has become the pursuit of surgeons. Based on renal cell carcinoma resection combined with zero ischemia technique, renal parenchyma, and renal function can be protected to the maximum extent on the premise of ensuring tumor safety.

The purpose of this study is to explore the safety and efficacy of zero-ischemia TE by analyzing the data of early renal cell carcinoma patients who had undergone PN and zero-ischemia TE before.

DETAILED DESCRIPTION:
According to the inclusion and exclusion criteria，collecting the data of participants who have undergone partial nephrectomy or renal tumor enucleation.

The investigators will compare the difference between TE and PN, clamped-enucleation and unclamped-enucleation, suture and sutureless zero-ischemia enucleation by the data the investigators collected.

After analysing the data, the investigators will discuss the safety and efficay of the sutureless zero-ischemia tumor enucleation. The patient who would be benefited from this operation and the patient who would be suggested to undergo this operation will also be discussed.

ELIGIBILITY:
Inclusion Criteria:

* 1. The age is between 18 and 80 years old.
* 2. Patients with T1a or T1b renal cell carcinoma according to TNM staging of AJCC renal cell carcinoma, 8th edition, 2017.
* 3. Patients who underwent unclamped renal tumor enucleation or partial nephrectomy between 2014 and 2022.

Exclusion Criteria:

* 1. The patients accompanied by severe active infection or severe diseases of heart, liver, kidney and hematopoietic system. And with other conditions that are not suitable for related tests.
* 2. The patient has no measurable or evaluable lesions.
* 3. The tumor is close to the collection system and touches the renal artery or renal vein. And other anatomy of tumor is not suitable for tumor enucleation.
* 4. History of organ transplantation or need long-term adrenocortical hormone therapy. Hypothyroidism, adrenal or pituitary dysfunction that cannot be controlled by hormone replacement therapy alone. type I diabetes mellitus, psoriasis or vitiligo that require systematic treatment, etc.
* 5. Active infection requiring systemic treatment. Human immunodeficiency virus (HIV) infection (known HIV antibody positive). Active HBV or HCV infection (HBsAg positive, or HBcAb positive but HBsAg negative, additional testing is required Quantitative DNA, the result does not exceed the upper limit of the laboratory normal value of the research center can participate in this study; the HCV RNA test result of the previous HCV infection screening period is negative, can participate in this study)
* 6. Patients have history of kidney surgery or any history of kidney inflammation surgery. Patients have kidney cancer related to urinary collection system and have other kidney diseases (including kidney stone glomerulonephritis)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with early renal carcinoma who have undergone partial nephrectomy or tumor enucleation.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Operation time | Period of surgery
  Operation time
Estimated blood loss | Period of surgery
  The estimated blood loss of operation
Positive rate of incision margin | Period of surgery
  Positive rate of incision margin
Serum creatinine | Pre-operative, 1 day after the surgery and monthly follow-up in one year
  Serum creatinine of patients before and after operation and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yichun Zheng, Doctor, Study Chair — The Fourth Affiliated Hospital Zhejiang University School of Medicine
Locations (1):
- The Fourth Affiliated Hospital Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu X, Chen W, Huang J, Zhang J, Liu D, Huang Y, Chen Y, Xue W. Zero ischemia laparoscopic microwave ablation assisted enucleation vs. laparoscopic partial nephrectomy in clinical T1a renal tumor: a randomized clinical trial. Transl Cancer Res. 2020 Jan;9(1):194-202. doi: 10.21037/tcr.2019.12.73. PMID 35117173
- [Derived] Xu C, Jiang Y, Du J, Yang K, Zhong Q, Liu D, Zhang C, Zheng Y. Three-dimensional reconstruction-guided modified arterial-based complexity scoring system for nephron-sparing surgery: comparative outcomes of on-clamp and off-clamp tumor enucleation in renal cell carcinoma. Front Surg. 2025 Nov 6;12:1683222. doi: 10.3389/fsurg.2025.1683222. eCollection 2025. PMID 41282560

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT05790122/Prot_SAP_000.pdf